CLINICAL TRIAL: NCT05244525
Title: Subacromial Injection of Epinephrine Improves Visualization in Shoulder Arthroscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, James M. Gregory, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSC-MS-21-1061
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Results first posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-10

CONDITIONS: Shoulder Arthroscopy
Keywords: Shoulder; Rotator Cuff; Epinephrine; Subacromial bursa
MeSH Terms: interventions — Bupivacaine; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Drug: Bupivacaine with Epinephrine
- Control Group (Active Comparator)
  Interventions: Drug: Bupivacaine alone

INTERVENTIONS:
Drug: Bupivacaine with Epinephrine — Randomization will be performed prior to surgery and group designation will be placed within an opaque envelope in the patient's chart.The circulating nurse will prepare the pre-operative injection. Study patients will receive an injection containing a total volume of 20 mL of bupivacaine with epinephrine (0.3 mL epinephrine in 30 mL of 0.5% bupivacaine).The syringe will not be labeled, and the contents of the injection will not be disclosed to the surgeon to preserve blinding. The injection will be performed with an 18-gauge needle into the subacromial space via a posterior or lateral approach after positioning the patient in the beach chair position, but prior to prepping and draping.Throughout the case, the mean arterial pressure of the patient will be monitored. At the conclusion of the surgical procedure, the surgeon will rate visual clarity on a visual analog scale. Changes in pump pressure from the initial pressure of 35mmHg during the surgical procedure will also be recorded.
  Arms: Treatment
Drug: Bupivacaine alone — Randomization will be performed prior to surgery and group designation will be placed within an opaque envelope in the patient's chart.The circulating nurse will prepare the pre-operative injection. Control patients will receive an injection containing 20mL of 0.5% bupivacaine alone.Throughout the case, the mean arterial pressure of the patient will be monitored. At the conclusion of the surgical procedure, the surgeon will rate visual clarity on a visual analog scale.Changes in pump pressure from the initial pressure of 35mmHg during the surgical procedure will also be recorded.
  Arms: Control Group

SUMMARY:
The purpose of this study is to evaluate surgeon-rated visual clarity and the need for increased irrigation pump pressure during arthroscopic shoulder surgery and to evaluate mean arterial pressure, operative time, and any adverse events that occur during arthroscopic shoulder surgery.

ELIGIBILITY:
Inclusion Criteria:

* Undergo arthroscopic shoulder surgery in the seated upright (beach-chair) position requiring visualization within the subacromial space

Exclusion Criteria:

* Are unable to provide informed consent
* Non-English speaker
* Have a history of adverse medication reaction to epinephrine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Gregory, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Feinstein S, Svetgoff RA, Harmon J, Siahaan J, Ngo DH, Fullick RK, Flores SE, Shupe PG, Gregory BP, Gregory JM. Effect of a Preoperative Subacromial Epinephrine Injection on Visualization During Shoulder Arthroscopic Surgery: A Randomized Controlled Trial. Orthop J Sports Med. 2024 Oct 10;12(10):23259671241278247. doi: 10.1177/23259671241278247. eCollection 2024 Oct. PMID 39399770

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Control Group
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Control Group | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 26 | 49
  >=65 years | 7 | 4 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 16 | 28
  Male | 18 | 14 | 32
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Surgeon-rated Visual Clarity as Assessed by the Visual Analog Scale
Description: This scale is scored from 1-10, a higher number indicating better clarity
Time Frame: end of surgery(about 30-120 minutes from start of surgery)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 30 | 30
score on a scale | 8.3 (1.4) | 7.5 (1.8)

2. Primary Outcome: Percentage of Participants for Whom Intra-operative Arthroscopic Pump Pressure Was Increased to 45mmHg or Higher During the Surgical Procedure
Description: The pump pressure is initially set at 35mmHg during the arthroscopic surgical procedure. If visualization is limited during the procedure, surgeons may increase the pump pressure of arthroscopic fluid within the shoulder during the procedure. This outcome measure reports the percentage of participants for whom intra-operative arthroscopic pump pressure was increased to 45mmHg or higher during the surgical procedure.
Time Frame: From start of surgery to end of surgery(about 30-120 minutes)
Measure: Number; unit: percent
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 30 | 30
percent | 22 | 23

3. Secondary Outcome: Intraoperative Mean Arterial Pressure
Time Frame: end of surgery(about 30-120 minutes from start of surgery)
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 30 | 30
mmHg | 70.5 (12.7) | 71.3 (7.3)

4. Secondary Outcome: Total Operative Time
Time Frame: end of surgery(about 30-120 minutes from start of surgery)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 30 | 30
minutes | 62 (19.4) | 64 (30.1)

5. Secondary Outcome: Number of Subjects Who Experience Intraoperative Adverse Events
Time Frame: end of surgery(about 30-120 minutes from start of surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

6. Secondary Outcome: Number of Subjects Who Experience Post Operative Adverse Events
Time Frame: from the end of surgery up to 2 weeks post surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment | Control Group
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: from start of surgery up to 2 weeks post surgery
Arm/Group | Treatment | Control Group
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-02): https://cdn.clinicaltrials.gov/large-docs/25/NCT05244525/Prot_SAP_000.pdf